CLINICAL TRIAL: NCT06585124
Title: Observational Study on the Application of Flow Cytometry for the Study of T-Cell Populations in Lymphoma-associated Hemophagocytic Lymphohistiocytosis
Brief Title: Flow Cytometry for the Study of T-Cell Populations in Hemophagocytic Lymphohistiocytosis Associated With Lymphomas
Acronym: LA-HLH
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ID-6536
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-07

CONDITIONS: Lymphoma; Hemophagocytic Lymphohistiocytoses
Keywords: Flow Cytometry; T cell activation; lymphoma; HLH
MeSH Terms: conditions — Lymphoma; Lymphohistiocytosis, Hemophagocytic | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Flow Cytometry — Study of t cell population in flow cytometry

SUMMARY:
The goal of this study is to explore the associations between T cell activation and the occurrence of hemophagocytic lymphohistiocytosis (HLH) in patients with newly diagnosed lymphomas. The specific aims are:

Prediction of Lymphoma-Associated HLH (LA-HLH): Compare flow cytometric T cell activation markers with the H-score to predict LA-HLH.

Identification of new markers for predicting HLH in patients with aggressive lymphoma.

Description of the incidence rate of LA-HLH. Assessment of the outcomes of LA-HLH identified by flow cytometric analysis or the H-score.

This prospective, single-center observational study will include 150 patients newly diagnosed with aggressive lymphoma within one year. Peripheral blood samples will be taken at diagnosis alongside routine blood chemistry tests for flow cytometric analysis of the T-lymphocyte activation profile. Data on disease characteristics will be collected to calculate the H-score, HLH-2004 score, and OHI score for diagnosing HLH. The flow cytometry results will be compared with these scores to evaluate their effectiveness in diagnosing LA-HLH.

DETAILED DESCRIPTION:
Hemophagocytic lymphohistiocytosis (HLH) is a rare and severe syndrome characterized by excessive immune system activation and dysregulation. This leads to an overproduction of cytokines and activation of the histiocytic-macrophage system, potentially resulting in multi-organ failure and death. HLH can be classified into primary and secondary forms. Secondary HLH is often triggered by infections, autoimmune diseases, or neoplasms, with lymphomas being the most frequent neoplastic triggers.

There is limited knowledge about secondary HLH, particularly regarding early diagnosis and optimal management. This project aims to address this gap by analyzing cytotoxic T-cells and cell expression markers using flow cytometry, building on findings from two pediatric studies.

Aggressive onset lymphomas may induce a systemic hyperinflammatory state, complicating the diagnosis of HLH, especially in the presence of concurrent bacterial or viral infections. Given the rarity of HLH and its poor prognosis if not promptly diagnosed, further research is crucial, especially in lymphoma-associated cases.

This study aims to apply T-cell activation profiling, previously demonstrated in pediatric populations, to patients with aggressive Non-Hodgkin's Lymphoma and Hodgkin's Lymphoma to identify HLH-associated cases at onset.

The study aims to include 150 patients diagnosed with aggressive lymphoma within a one-year period A peripheral blood sample, collected alongside routine blood chemistry tests at diagnosis, will be used for the flow cytometric study of the T-lymphocyte activation profile. Data pertaining to disease characteristics will be gathered to calculate diagnostic scores for HLH, including the H-score, HLH-2004 score, and OHI score. The flow cytometry results will then be compared with these score parameters to assess their correlation with the diagnosis of lymphoma-associated HLH (LA-HLH).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Diagnosis at onset of aggressive lymphoma including the following histotypes:

   * Hodgkin lymphoma
   * Transformed B cell lymphomas;
   * Diffuse large B-cell lymphomas (diffuse large B-cell lymphoma NOS; T-cell/histiocyte-rich B-cell lymphoma; High grade B-cell lymphoma/high grade B-cell lymphoma with MYC and BCL2 rearrangement ALK-positive large B-cell lymphoma; Large B-cell lymphoma with IRF4 rearrangement; High grade B-cell lymphoma with 11q alterations; Lymphomatoid granulomatosis; EBV-positive large B-cell lymphoma Large B-cell lymphoma associated with chronic inflammation; Fibrin-associated large B-cell lymphoma; Fluid overload-associated large B-cell lymphoma; Plasmoblastic lymphoma; Immune-privileged site B-cell lymphoma Primary cutaneous leg-type large B-cell lymphoma; Intravascular large B-cell lymphoma; Primary mediastinal large B-cell lymphoma; Mediastinal grey zone lymphoma; High grade NOS B-cell lymphoma)
   * Burkitt lymphoma
   * KSHV/HHV8 a ssociatedlymphomas
   * Lymphomas associated with immunodeficiency or immune dysregulation
   * Mature T-cell-derived lymphomas (NOS peripheral T-cell lymphoma; Nodal follicular helper T-cell lymphoma; Anaplastic large cell lymphoma; Nodal and extranodal EBV-positive T/NK-cell lymphomas; Hepatosplenic T-cell lymphoma; Enteropathy-associated intestinal T-cell lymphoma, epitheliotropic monomorphic and NOS; Subcutaneous T-cell lymphoma similar to panniculitis)
3. Informed consent to the use of biologic materials for studies related to the present proposal.

Exclusion Criteria:

1. Diagnosis of indolent non-Hodgkin's lymphoma or diagnoses other than those listed in the inclusion criteria
2. Prolonged steroid therapy, defined as lasting more than 15 days or high doses of steroid, exceeding 1 mg/kg
3. Age ≤ 18 years;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with newly diagnosed lymphomas
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Assocation of flow cytometry parameters on peripheral blood with the H-score, the standard for the diagnosis of lymphoma-associated HLH | 2 years
  Diagnostic rate of flow cytometry for lymphoma-associated HLH

SECONDARY OUTCOMES:
Determine the incidence of LA-HLH | 2 years
  incidence rate
To evaluate the outcome of patients with LA-HLH | 2 years
  overall survival
Define the rate of complete responses to lymphoma treatment | 2 years
  Complete remission rate

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Hohaus, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Stefan Hohaus, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Decision on IPD will be jointly made by investigators at end of study